CLINICAL TRIAL: NCT05850195
Title: Assessment Of Different Indices in Prediction of Noninvasive Ventilation Failure in Patients With Acute Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Abd El Razek Kamel, lecturer assistant, Assiut University
Other Study IDs: NIV failure in acute RF
Record Dates: First submitted 2023-03-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Non-invasive Ventilation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Other: non invasive ventilation — compare indices and diaphragmatic ultrasonography for prediction of NIV failure in acute RF patients

SUMMARY:
This study will use different indices for prediction of NIV failure in ARF patients Evaluation of HACOR score and ROX index for early prediction of NIV failure in patients with ARF.

Study value of diaphragmatic dysfunction assessed by ultrasound as tool for prediction of success of NIV in ARF patients.

Compare clinical significance of these scoring systems between hypoxemic and hypercapnic RF

DETAILED DESCRIPTION:
Noninvasive ventilation (NIV) is a useful and safe method to improve gas exchange in patients with acute respiratory failure (ARF) of different etiologies. NIV reduces the work of breathing, improves arterial oxygenation and alveolar ventilation. It is associated with improved survival in the acute care setting (Cabrini L 2015) when compared to conventional oxygen therapy. As NIV offers several major advantages over invasive ventilation (e.g., preserving the ability to swallow, cough, and communicate verbally), it is widely used to avoid intubation.

Although NIV nowadays is frequently used, its failure rate remains high (25-59%), indicating that not all patients benefit from this treatment. There is an association between the unsuccessful NIV and the poor outcome has been suggested. Among patients who experience NIV failure, either premature or delayed NIV discontinuation further increases mortality. Thus, identifying the predictors of NIV failure is crucial because of the strong link between failure and poor outcomes. So, researchers woke to make scoring systems that may predict NIV failure, as HACOR and ROX indices.

Recently, ultrasonography (US) of the diaphragm as a bedside method is used for evaluation of diaphragmatic function and predicting failure of NIV in acutely ill patients.

Up till now there is limited research to support significance of different indices for prediction of NIV failure and need for invasive mechanical ventilation (IMV).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute hypoxic respiratory failure who need Noninvasive ventilation.
2. Patients with acute hypercapnic respiratory failure who need Noninvasive ventilation.

Exclusion Criteria:

1. Age < 18 years old.
2. Patients with unconsciousness, severe hemodynamic instability, unable to fit mask (Recent facial surgery, trauma, or deformity), inability to protect the airway or clear respiratory secretions or any other contraindication of NIV.
3. neuromuscular disease or chest wall deformities.
4. Pregnancy.
5. NIV intolerance.
6. severe obesity with Body Mass Index (BMI)≥35 kg/m2

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of both gender with acute respiratory failure either hypoxic or hypercapnic who need Noninvasive ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
measure value of HACOR score for prediction of failure of NIV in ARF patients. | Baseline (before starting NIV treatment)
  HACOR score (Heart rate, Acidosis, Consciousness, Oxygenation, Respiratory rate) It will be analyzed as continuous value and dichotomized as ≤ or > 5
measure value of HACOR score for prediction of failure of NIV in ARF patients. | at 1 hour of NIV treatment
  HACOR score (Heart rate, Acidosis, Consciousness, Oxygenation, Respiratory rate) It will be analyzed as continuous value and dichotomized as ≤ or > 5
measure value of HACOR score for prediction of failure of NIV in ARF patients. | at 6 hours of NIV treatment
  HACOR score (Heart rate, Acidosis, Consciousness, Oxygenation, Respiratory rate) It will be analyzed as continuous value and dichotomized as ≤ or > 5
measure value of HACOR score for prediction of failure of NIV in ARF patients. | at 12 hours of NIV treatment
  HACOR score (Heart rate, Acidosis, Consciousness, Oxygenation, Respiratory rate) It will be analyzed as continuous value and dichotomized as ≤ or > 5
measure value of HACOR score for prediction of failure of NIV in ARF patients. | at 24 hours of NIV treatment
  HACOR score (Heart rate, Acidosis, Consciousness, Oxygenation, Respiratory rate) It will be analyzed as continuous value and dichotomized as ≤ or > 5
measure value of HACOR score for prediction of failure of NIV in ARF patients. | at 48 hours of NIV treatment
  HACOR score (Heart rate, Acidosis, Consciousness, Oxygenation, Respiratory rate) It will be analyzed as continuous value and dichotomized as ≤ or > 5
measure value of ROX index for prediction of failure of NIV in ARF patients. | Baseline (before starting NIV treatment)
  ROX index is the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ fraction of inspired oxygen (FIO2) to respiratory rate (RR). It will be analyzed as continuous value and dichotomized as < or ≥ 4.88
measure value of ROX index for prediction of failure of NIV in ARF patients. | at first hour of NIV treatment
  ROX index is the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ fraction of inspired oxygen (FIO2) to respiratory rate (RR). It will be analyzed as continuous value and dichotomized as < or ≥ 4.88
measure value of ROX index for prediction of failure of NIV in ARF patients. | at 6 hours of NIV treatment
  ROX index is the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ fraction of inspired oxygen (FIO2) to respiratory rate (RR). It will be analyzed as continuous value and dichotomized as < or ≥ 4.88
measure value of ROX index for prediction of failure of NIV in ARF patients. | at 12 hours of NIV treatment
  ROX index is the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ fraction of inspired oxygen (FIO2) to respiratory rate (RR). It will be analyzed as continuous value and dichotomized as < or ≥ 4.88
measure value of ROX index for prediction of failure of NIV in ARF patients. | at 24 hours of NIV treatment
  ROX index is the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ fraction of inspired oxygen (FIO2) to respiratory rate (RR). It will be analyzed as continuous value and dichotomized as < or ≥ 4.88
measure value of ROX index for prediction of failure of NIV in ARF patients. | at 48 hours of NIV treatment
  ROX index is the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ fraction of inspired oxygen (FIO2) to respiratory rate (RR). It will be analyzed as continuous value and dichotomized as < or ≥ 4.88
diaphragmatic thickness assessment by ultrasound | at first 1 day of starting NIV treatment
  ultrasonographic measurement of diaphragmatic thickness fraction for prediction of failure of NIV in ARF patients.
diaphragmatic dysfunction assessment by ultrasound | at first 1 day of starting NIV treatment
  ultrasonographic measurement of diaphragmatic excursion for prediction of failure of NIV in ARF patients.

REFERENCES:
- [Background] Demoule A, Girou E, Richard JC, Taille S, Brochard L. Benefits and risks of success or failure of noninvasive ventilation. Intensive Care Med. 2006 Nov;32(11):1756-65. doi: 10.1007/s00134-006-0324-1. Epub 2006 Sep 21. PMID 17019559
- [Background] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830